CLINICAL TRIAL: NCT01208610
Title: The Effectiveness of Adopting Humanized Service Program on Transabdominal Ultrasound About Pregnant Women's Service Quality and Satisfaction
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ya-Ling Wu, Department of Obsterics and Gynecology
Other Study IDs: 99015
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Pregnant Women

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Effectiveness of Adopting Humanized Service Program on Transabdominal Ultrasound About Pregnant Women's Service Quality and Satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. Adult over the age of 20 pregnant women.
2. Clear consciousness, those without severe cognitive impairment, such as dementia, mental retardation or mental illness.
3. Literacy and the use of Chinese or Taiwanese.
4. Willingness to participate in the research.

Exclusion Criteria:

Refused to participate in the research

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-02; Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Wu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan